CLINICAL TRIAL: NCT01712451
Title: Dose-ranging Study of the Safety and Efficacy of Fluticasone Propionate and Salmeterol Xinafoate in Healthy Patients With Abdominal Contour Defects
Brief Title: Dose-ranging Study
Acronym: LIPO-102-CL-11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPO-102-CL-11
Record Dates: First submitted 2012-10-16; First posted 2012-10-23 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Abdominal Contour Defects
Keywords: adiposity
MeSH Terms: conditions — Obesity | interventions — Fluticasone-Salmeterol Drug Combination; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- LIPO-102, Low (Experimental)
  Interventions: Drug: salmeterol xinafoate, fluticasone propionate
- LIPO-102, Mid (Experimental)
  Interventions: Drug: salmeterol xinafoate, fluticasone propionate
- LIPO-102, High (Experimental)
  Interventions: Drug: salmeterol xinafoate, fluticasone propionate
- LIPO-102; Placebo (Experimental)
  Interventions: Drug: Placebo
- salmeterol xinafoate (Experimental)
  Interventions: Drug: salmeterol xinafoate

INTERVENTIONS:
Drug: salmeterol xinafoate, fluticasone propionate — LIPO-102
  Other Names: LIPO-102
  Arms: LIPO-102, High; LIPO-102, Low; LIPO-102, Mid
Drug: Placebo — Placebo
  Arms: LIPO-102; Placebo
Drug: salmeterol xinafoate — Salmeterol
  Arms: salmeterol xinafoate

SUMMARY:
Dose ranging study

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years of age inclusive
* abdominal contour defect
* BMI <25 kg/msq
* Stable diet and exercise and body weight

Exclusion Criteria:

* Prior treatment of abdominal contour defects (liposuction, abdominoplasty, etc)
* Known hypersensitivity to study drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety | 8 weeks treatment
  physical exam, vital signs, clinical assessment of injection, clinical laboratory tests, and adverse events
Change in abdominal circumference | Baseline to 9 weeks
  abdominal circumference

SECONDARY OUTCOMES:
Change in global clinician scale score | Baseline to 9 weeks
Change in global patient scale score | Baseline to 9 weeks
Change in Photonumeric scale score | Baseline to 9 weeks
Change in Patient Reported Outcome Score | Baseline to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murray Maytom, Study Director — Neothetics, Inc
Locations (6):
- United States (6):
  - Beverly Hills, California
  - San Diego, California
  - New York, New York
  - Raleigh, North Carolina
  - Nashville, Tennessee
  - Plano, Texas